CLINICAL TRIAL: NCT00842517
Title: A Behavioral Model for Maintenance of Drug Abstinence
Brief Title: Long Term Maintenance of Drug Abstinence
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Treatment Research Institute (Other)
Responsible Party: Kimberly C. Kirby, Ph.D., Treatment Research Institute
Organization: Public Health Management Corporation (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0308; R01DA017444 (NIH)
Record Dates: First submitted 2007-10-24; First posted 2009-02-12 (Estimated); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Cocaine Dependence; Cocaine Abuse
Keywords: Cocaine Dependence; Cocaine Abuse; Substance Abuse; Contingency Management; Drug Treatment
MeSH Terms: conditions — Cocaine-Related Disorders; Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Extended (Experimental): 36-week duration contingency management program
  Interventions: Behavioral: Contingency Management
- Standard (Active Comparator): 12-week duration contingency management program
  Interventions: Behavioral: Contingency Management

INTERVENTIONS:
Behavioral: Contingency Management

SUMMARY:
The purpose of this study is to develop a model for long-term maintenance of behavior change by examining the effects of extending the duration of contingency management (CM) for drug abuse on long-term abstinence outcomes. The primary hypothesis is that the Extended (36 week) CM group will have better long-term outcomes as exhibited by greater rates of abstinence at each follow-up assessment as compared to the Standard (12 week) CM group.

DETAILED DESCRIPTION:
This protocol examines the effects of extending the duration of contingency management (CM) for drug abuse and dependence on long-term abstinence outcomes. Following the tenets of basic behavioral research, we have outlined a model for long-term behavior maintenance that suggests that successful long-term behavior change does not focus on undoing old behaviors, but concentrates on developing new behaviors in a wide variety of new contexts, and provides enduring reinforcement for the new behaviors. The implication of this model is that in order to develop strategies for supporting long-term behavior change we need to determine the optimal duration of continuing treatment-arranged contingencies, better specify incompatible behaviors that emerge for patients who are successful in sustaining periods of continuous drug abstinence, and determine which incompatible behaviors are most likely to have naturally-occurring sustaining contingencies of reinforcement. This research will examine the model by randomly assigning cocaine-dependent or cocaine-abusing methadone maintenance patients to either a Standard (12 week) or Extended (36 week) period of contrived contingencies. We will be conducting a 2 year follow-up in order to investigate whether providing a longer duration of CM will result in a greater proportion of abstinent individuals during this time, how long the abstinence will last and to discover if longer durations of drug abstinence during the first year after treatment entry will predict better longer-term abstinence outcomes. We also compare outcomes on abstinence-related behaviors to see if provision of an extended voucher program leads to an increase in non-drug using natural reinforcers and activities. This study participates in the NIH-sponsored Health Maintenance Consortium designed to promote interchange of concepts, methods and measures related to the maintenance of long-term behavior change.

ELIGIBILITY:
Inclusion Criteria:

* Meet DSM-IV criteria for current cocaine dependence or abuse
* Be willing and able to give valid contact information
* Be receiving a stable dose of 40 milligrams or more of methadone

Exclusion Criteria:

* Are unable to give informed consent (fails simple open-ended consent quiz)
* Answer yes to the question "Are you in recovery from gambling? That is, have you stopped gambling because of previous problems with gambling?"
* Report that they have a romantic partner who is already participating in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2004-09; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Duration of cocaine abstinence | Every 2 weeks for the first year the participant is involved in the study; in addition to 3 month, 6 month, 9 month, 12 month, 15 month, 18 month, 21 month, and 24 month assessment points.

SECONDARY OUTCOMES:
The presence and frequency of non-drug using activities | 3 month, 6 month, 9 month, 12 month, 15 month, 18 month, 21 month, 24 month
The presence and frequency of natural contingencies of reinforcement | 3 month, 6 month, 9 month, 12 month, 15 month, 18 month, 21 month, 24 month
The presence and frequency of meaningful correlates of long-term behavior change | Every 2 weeks for the first year the participant is involved in the study; in addition to 3 month, 6 month, 9 month, 12 month, 15 month, 18 month, 21 month, and 24 month assessment points.

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly C Kirby, Ph.D., Principal Investigator — Treatment Research Institute
Locations (1):
- Parkside Recovery, Philadelphia, Pennsylvania, United States